CLINICAL TRIAL: NCT00098163
Title: A Phase I Study to Evaluate the Safety and Immunogenicity of ALVAC-HIV vCP1521 in Infants Born to HIV-1 Infected Women in Uganda
Brief Title: Safety of and Immune Response to an HIV-1 Vaccine (ALVAC-HIV vCP1521) in Infants Born to HIV Infected Mothers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPTN 027; 10141 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: ALVAC-HIV vCP1521
- 2 (Placebo Comparator)
  Interventions: Biological: ALVAC HIV-1 vCP1521

INTERVENTIONS:
Biological: ALVAC-HIV vCP1521 — One 1-ml dose of HIV-1 vaccine administered after birth on or before Day 3 and at weeks 4, 8, and 12.
  Arms: 1
Biological: ALVAC HIV-1 vCP1521 — One 1-ml dose of HIV-1 vaccine placebo administered after birth on or before Day 3 and at Weeks 4, 8, and 12.
  Arms: 2

SUMMARY:
The purpose of this study is to test the safety of and immune response to an HIV-1 vaccine, ALVAC-HIV vCP1521, given to infants born to HIV-1 infected mothers in Uganda.

DETAILED DESCRIPTION:
Mother-to-child transmission (MTCT) of HIV can be caused either by perinatal transmission of HIV or by breastfeeding, a common practice in poorer regions of the world. HIV preventive vaccines are currently under investigation as potential solutions to worldwide MTCT of HIV. This study will evaluate the safety and immunogenicity of an HIV-1 vaccine, ALVAC-HIV vCP1521, in infants born to HIV-1 infected mothers in Uganda. The vaccine is a preparation of a live attenuated recombinant canarypox virus, encoding HIV clades B and E envelope proteins. This study will be conducted at Mulago Hospital in Uganda.

Mothers will enroll in this study during their third trimesters of pregnancy. During screening, mothers will undergo medical history assessment, a physical exam, and blood collection. After delivery and prior to infant enrollment, mothers will have another physical exam; mothers and their infants will be accompanied home by a home visitor who will document contact information.

Infants will be followed for 24 months after birth. Infants will be randomly assigned to receive 4 injections of vaccine or placebo. Study injections will be given at the start of the study and at Weeks 4, 8, and 12. Infants will be observed for 1 hour after each vaccine administration to check for body temperature and local and systemic reactions. They will also be evaluated in the clinic the day after each immunization for any local or systemic reactions. Infants will be visited at home 2 days after vaccine administration by a trained study nurse who will assess reactogenicity. Blood will be collected at 9 selected times: study entry, Weeks 2, 6, 10, and 14, and Months 6, 12, 18, and 24. Sixteen study visits occurring over 2 years will include medical history assessment and physical exams. Childhood immunizations will be given to infants at study entry and at Weeks 6, 10, and 14 and Months 6 and 12.

ELIGIBILITY:
Inclusion Criteria for HIV Infected Women:

* HIV infected
* In third trimester of pregnancy
* CD4 count of more than 500 cells/mm3 at screening
* Intends to give birth at Mulago Hospital, Uganda
* Willing to be taken home by a home visitor after delivery to document locator information and willing to be visited at home later

Inclusion Criteria for Infants Born to HIV Infected Women:

* 3 or fewer days of age
* Born to an HIV infected woman eligible for the study
* Weight at birth at least 2000 g (4.4 lbs)

Exclusion Criteria for HIV Infected Women:

* Prior participation in an HIV-1 vaccine trial
* Investigational agents, blood products, immunoglobulin, or immunotherapy any time during this pregnancy
* Documented or suspected serious medical illness or life-threatening condition that may interfere with the study
* Multiple birth predicted in current pregnancy

Exclusion Criteria for Infants Born to HIV Infected Women:

* Mother left study prior to infant enrollment and randomization
* Mother or infant received any active or passive HIV immunotherapy or investigational product other than the study vaccine. Mothers and infants who have taken nevirapine prior to study entry are not excluded.
* Blood products, immunoglobulin, or immunosuppressive therapy during labor and delivery or prior to study enrollment
* Abnormal vital signs prior to vaccination or clinical symptoms that may interfere with vaccine reaction assessment
* Part of a multiple birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Grade 3 or higher adverse events attributable to the vaccine. Mild and moderate adverse event rates will also be tabulated | At Day 0 and throughout study
Cell-mediated immunologic response as measured by HIV-specific cytotoxic T-lymphocyte activity against viral antigens | At Day 0 and throughout study
Humoral immunologic response as measured by detection of binding antibody to vaccine antigens and by neutralizing antibody assay | At Day 0 and throughout study

SECONDARY OUTCOMES:
Immune status as measured by CD4 cell counts in all immunized infants | Over the 24-month follow-up period
Development of immunity to routine vaccination as measured by antibody levels and Bacillus Calmette-Guéerin (BCG) scar formation | At the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Laura Guay, MD, Study Chair — Department of Pathology, Johns Hopkins University; Francis Mmiro, MBChB, FRCOG, Study Chair — Department of Obstetrics and Gynecology, Makerere University
Locations (1):
- Makerere University- JHU Research Collaboration {MUJHU CARE LTD} CRS, Kampala, Uganda

REFERENCES:
- [Background] Cao H, Mani I, Vincent R, Mugerwa R, Mugyenyi P, Kanki P, Ellner J, Walker BD. Cellular immunity to human immunodeficiency virus type 1 (HIV-1) clades: relevance to HIV-1 vaccine trials in Uganda. J Infect Dis. 2000 Nov;182(5):1350-6. doi: 10.1086/315868. Epub 2000 Oct 9. PMID 11023458
- [Background] de Bruyn G, Rossini AJ, Chiu YL, Holman D, Elizaga ML, Frey SE, Burke D, Evans TG, Corey L, Keefer MC. Safety profile of recombinant canarypox HIV vaccines. Vaccine. 2004 Jan 26;22(5-6):704-13. doi: 10.1016/j.vaccine.2003.08.023. PMID 14741163
- [Background] Franchini G, Gurunathan S, Baglyos L, Plotkin S, Tartaglia J. Poxvirus-based vaccine candidates for HIV: two decades of experience with special emphasis on canarypox vectors. Expert Rev Vaccines. 2004 Aug;3(4 Suppl):S75-88. doi: 10.1586/14760584.3.4.s75. PMID 15285707
- [Background] Safrit JT, Ruprecht R, Ferrantelli F, Xu W, Kitabwalla M, Van Rompay K, Marthas M, Haigwood N, Mascola JR, Luzuriaga K, Jones SA, Mathieson BJ, Newell ML; Ghent IAS Working Group on HIV in Women Children. Immunoprophylaxis to prevent mother-to-child transmission of HIV-1. J Acquir Immune Defic Syndr. 2004 Feb 1;35(2):169-77. doi: 10.1097/00126334-200402010-00012. PMID 14722451
- [Derived] Kaleebu P, Njai HF, Wang L, Jones N, Ssewanyana I, Richardson P, Kintu K, Emel L, Musoke P, Fowler MG, Ou SS, Jackson JB, Guay L, Andrew P, Baglyos L, Cao H; HPTN 027 protocol team. Immunogenicity of ALVAC-HIV vCP1521 in infants of HIV-1-infected women in Uganda (HPTN 027): the first pediatric HIV vaccine trial in Africa. J Acquir Immune Defic Syndr. 2014 Mar 1;65(3):268-77. doi: 10.1097/01.qai.0000435600.65845.31. PMID 24091694
- [Derived] Kintu K, Andrew P, Musoke P, Richardson P, Asiimwe-Kateera B, Nakyanzi T, Wang L, Fowler MG, Emel L, Ou SS, Baglyos L, Gurunathan S, Zwerski S, Jackson JB, Guay L. Feasibility and safety of ALVAC-HIV vCP1521 vaccine in HIV-exposed infants in Uganda: results from the first HIV vaccine trial in infants in Africa. J Acquir Immune Defic Syndr. 2013 May 1;63(1):1-8. doi: 10.1097/QAI.0b013e31827f1c2d. PMID 23221981